CLINICAL TRIAL: NCT00647075
Title: A Randomized, Parallel, Double-blind, Placebo-controlled, Pilot Clinical Study on the Effects of Yunzhi as Dietary Supplement in 60 Adult Patients Undergoing Adjuvant/Neoadjuvant Chemotherapy for Breast Cancer.
Brief Title: Yunzhi as Dietary Supplement in Breast Cancer
Acronym: YUNZHI-BC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Vita Green Health Products Co. Ltd., Vita Green Europe, S.A.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YUNZHI-BC
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; undergoing; adjuvant/neoadjuvant chemotherapy; symptomatic therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Yunzhi extract 3.5 g/day
  Interventions: Dietary Supplement: Yunzhi extract
- 2 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Yunzhi extract — 3.5 g/day
  Arms: 1
Dietary Supplement: Placebo — Placebo (starch)
  Arms: 2

SUMMARY:
The purpose of this study is to assess the effects of a dietary supplement, the traditional Asian mushroom Yunzhi, as adjuvant in the treatment of patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women with diagnosis of breast cancer
2. Undergoing adjuvant/neoadjuvant chemotherapy with either FEC, FAC, TAC, or EC + docetaxel combinations.
3. ≥ 18 years of age
4. Performance status: 0-2
5. Ability to provide written informed consent

Exclusion Criteria:

1. Any prior history of yunzhi use
2. Use of other herbal remedies during the study duration
3. Significant cardiac, pulmonary, renal, hepatic, gastrointestinal, CNS, psychiatric disease or illicit substance use/abuse that in the opinion of the investigator would make the participant a poor candidate for study participation
4. Pregnancy (for women of childbearing potential, a negative pregnancy test, urine or serum, is required within 14 days prior to randomization)
5. Systemic use of progestins, androgens or other steroids (dexamethasone is allowed if used as antiemetic therapy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Mean change in signs and symptoms from baseline measured by Visual Analogue Scale (VAS) | 6 months

SECONDARY OUTCOMES:
Treatment adherence Clinical and laboratory (including RBC, WBC and platelets) adverse events Adherence to chemotherapy schedule EPO and blood transfusion needs | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pere Gascon, MD, Principal Investigator — Hospital Clinic
Locations (2):
- Spain (2):
  - Hospital Clinic, Barcelona, Barcelona
  - Hospital Parc Tauli, Sabadell, Barcelona